CLINICAL TRIAL: NCT03284346
Title: Circuit, Interval-Based Aerobic and Resistance Exercise to Target Metabolic Dysregulation: The CARE Study for Breast and Prostate Cancer Survivors
Brief Title: Exercise in Targeting Metabolic Dysregulation in Stage I-III Breast or Prostate Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0S-17-5; NCI-2017-01426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-17-5 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-08-19; First posted 2017-09-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cancer Survivor; No Evidence of Disease; Obesity; Overweight; Prostate Carcinoma; Sedentary Lifestyle; Stage I Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Obesity; Overweight; Prostatic Neoplasms; Sedentary Behavior; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (CARE) (Experimental): Patients undergo supervised exercise sessions comprised of CARE over 50 minutes 3 days weekly for 16 weeks. Patients receive a Polar heart rate monitor to monitor heart rate during the CARE sessions.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Polar heart rate monitor; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (standard stretching) (Active Comparator): Patients undergo a standard stretching program 3 days weekly for 16 weeks. After 16 weeks, patients may undergo supervised exercise sessions comprised of CARE as in Arm I.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo CARE
  Arms: Arm I (CARE)
Behavioral: Exercise Intervention — Undergo standard stretching program
  Arms: Arm II (standard stretching)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Polar heart rate monitor — Receive Polar heart rate monitor
  Other Names: Monitor
  Arms: Arm I (CARE)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies how well circuit, interval-based aerobic and resistance exercise works in targeting metabolic dysregulation in stage I-III breast or prostate cancer survivors. Circuit, interval-based aerobic and resistance exercise may help to improve cardiovascular fitness, weight loss, healthy lifestyle behaviors, and muscle strength in breast or prostate cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effects of a 4-month circuit, interval-based aerobic and resistance exercise (CARE) intervention on metabolic dysregulation.

SECONDARY OBJECTIVES:

I. To determine the effects of a 4-month CARE intervention on sarcopenic obesity.

TERTIARY OBJECTIVES:

I. To determine the effects of a 4-month CARE intervention on skeletal muscle strength, physical fitness, and quality of life (QOL).

II. To determine the effects of a 4-month CARE intervention on vascular function.

OUTLINE: Patients are randomized to 1 of 2 arms.

Arm I: Patients undergo supervised exercise sessions comprised of CARE over 50 minutes 3 days weekly for 16 weeks. Patients receive a Polar heart rate monitor to monitor heart rate during the CARE sessions.

Arm II: Patients undergo a standard stretching program 3 days weekly for 16 weeks. After 16 weeks, patients may undergo supervised exercise sessions comprised of CARE as in Arm I.

After completion of study, patients undergoing CARE are followed up for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* BREAST CANCER COHORT:
* Women newly diagnosed (stage I-III) breast cancer
* Are overweight or obese with the following criteria (determined by study team at eligibility screening): body mass index (BMI) > 25 kg/m^2 (calculated using height and weight; an upper limit BMI will not be set; we will rely on obtaining physicians? clearance to assess full eligibility) or body fat > 30% (estimated by bioelectrical impedance), and waist circumference > 35 in
* Have undergone a lumpectomy or mastectomy
* Have completed cancer-related treatment within the past 3 years
* Speak English or Spanish
* Are in breast cancer remission with no detectable disease present
* Able to initiate a supervised exercise program (free from any cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity)
* Free from history of chronic disease including uncontrolled diabetes (fasting blood glucose > 125 mg/dL), hypertension (blood pressure > 130/90 mmHg) or thyroid disease (< 0.4 or > 4.0 mIU/L); this will be determined by review of medical records and/or physician clearance
* Have not experienced a weight reduction >= 10% within past 6 months
* Currently participate in less than 60 minutes of structured exercise/week
* No planned reconstructive surgery with flap repair during trial and follow-up period
* May use adjuvant endocrine therapy if use will be continued for duration of study intervention
* Do not smoke (no smoking during previous 12 months)
* Willing to travel to the exercise facility at University of Southern California (USC)
* PROSTATE CANCER COHORT:
* Men > 18 diagnosed with prostate cancer for which antiandrogen therapy (ADT) (castration therapy) is being prescribed for at least 16 weeks; castration may be achieved surgically or using gonadotrophin releasing hormone (LHRH) agonists (i.e. leuprolide, goserelin, etc.) or LHRH antagonists (i.e. degarelix)
* Additional ADT agents may be concurrently administered (abiraterone, bicalutamide, enzalutamide, etc.)
* Men must be obese (BMI > 25) and sedentary (< 60 minutes of structured exercise per week)

Exclusion Criteria:

* Patients with metastatic disease (BREAST ONLY)
* Have not completed surgery, chemotherapy, or radiation treatment associated with their diagnosis; a washout period of a minimum of 6 weeks is required from the last anti-cancer treatment received except hormonal therapy
* Patients with a history of any musculoskeletal, cardiorespiratory or neurological diseases that preclude the participation in exercise must be evaluated by their physician to assess if they are suitable to proceed on study
* Are planning reconstructive surgery with flap repair during trial and follow-up period
* Are unable to travel to the exercise facility at USC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Change in insulin resistance | Baseline up to week 34
  Homeostasis Model Assessment (HOMA) will be used to estimate insulin resistance using fasting plasma levels of glucose and insulin.
Change in metabolic syndrome (Blood Pressure) | Baseline up to week 34
  Blood pressure will be measured using an automated device with an appropriate sized cuff (Omron BP 786, Lake Forest, IL) after the participant has sat quietly for 5 minutes while resting his/her arm on a table so the brachial artery is level with the heart.
Change in metabolic syndrome (Waist Circumference) | Baseline up to week 34
  A tape measure will be used to obtain waist circumference defined as the distance around the waist using the umbilicus as the reference point.
Change in metabolic syndrome (Fasting Plasma Levels of Glucose) | Baseline up to week 34
  The investigators will assess fasting plasma levels of glucose at baseline, weeks 9, 18 and 34.
Change in metabolic syndrome (High-Density Lipoprotein-Cholesterol) | Baseline up to week 34
  The investigators will assess high-density lipoprotein-cholesterol levels at baseline, weeks 9, 18 and 34.
Change in metabolic syndrome (Triglycerides) | Baseline up to week 34
  The investigators will assess triglyceride levels at baseline, weeks 9, 18 and 34.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States